CLINICAL TRIAL: NCT04845815
Title: Patterns of Renal Tubular Disorders in Egyptian Children: a Single Center Study
Brief Title: Renal Tubular Disorders in Egyptian Children
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ashraf Mohamed, Principal investigator and resident Doctor in Paediatric Department, Sohag University
Other Study IDs: Soh-Med-21-04-04
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2021-04

CONDITIONS: Renal Tubular Disorders in Children
Keywords: renal tubular disorders; failure to thrive; metabolic acidosis; metabolic alkalosis; hypokalemia
MeSH Terms: conditions — Failure to Thrive; Acidosis; Hypokalemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Renal tubules play an important role in fluid, electrolyte, and acid-base homeostasis. Defect of these functions can give rise to a host of disorders. These disorders can lead to life threatening disturbances in electrolytes and acid-base balance. In Egypt, there is little data about these disorders. Many of these cases are diagnosed late, therefore Early suspicion for diagnosis can improve the overall clinical outcome of these children.

DETAILED DESCRIPTION:
Renal tubules play an important role in fluid, electrolyte, and acid-base homeostasis. Defect of these functions can give rise to a host of disorders. These disorders can lead to life threatening disturbances in electrolytes and acid-base balance. In Egypt, there is little data about these disorders. Many of these cases are diagnosed late, therefore Early suspicion for diagnosis can improve the overall clinical outcome of these children. As a result, starting management early will help those children have a better life. Therefore awareness about these disorders and long-term outcome is really important. The investigators present the clinical characterizations of many tubular disorder and the follow up in our center.

The aim of this study is to reveal the different clinical presentations and the main lab features of renal tubular disorders in children to promote early recognition and management.

ELIGIBILITY:
Inclusion Criteria:

* All children aged from one month to 18 years who have renal tubular disorders.

Exclusion Criteria:

* Children who have renal tubular disorders secondary to drugs, intoxication, obstructive uropathy or transient in nature.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all children who have renal tubular disorders (inpatient and outpatient) in the Paediatric Department, Sohage University Hospital.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
weight | 1 years
  in kilograms
Glomerular function | 1 years
  The glomerular function was assessed by estimated glomerular filtration rate (eGFR) calculated using Schwartz formula. Chronic kidney disease (CKD) was defined in the presence of a permanent reduction in GFR (e-GFR; <60 ml/min/1.73 m2 Kidney Disease Outcomes Quality Initiative < stage 3).
height | 1 years
  in meters

CONTACTS AND LOCATIONS:
Locations (1):
- pediatric department, Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT04845815/Prot_SAP_000.pdf